CLINICAL TRIAL: NCT03196102
Title: Evaluation of a Brief Tobacco Intervention in the US Military
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Melissa Little, PhD, MPH, Associate Professor, Department of Public Health Sciences, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-04697-XP DoD
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Tobacco Use; Tobacco Smoking; Smoking, Cigar; Smoking, Pipe; Smoking, Hookah; Nicotine Dependence
Keywords: tobacco prevention; tobacco intervention; military; brief intervention
MeSH Terms: conditions — Tobacco Use; Tobacco Smoking; Cigar Smoking; Pipe Smoking; Water Pipe Smoking; Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BTI + Cigarette smoking military tailored pamphlet (Experimental): BTI + Cigarette smoking military tailored pamphlet
  Interventions: Behavioral: BTI; Behavioral: Cigarette smoking military tailored pamphlet
- Cigarette smoking military tailored pamphlet (Active Comparator): Cigarette smoking military tailored pamphlet
  Interventions: Behavioral: Cigarette smoking military tailored pamphlet
- Standard smoking cessation pamphlet (Active Comparator): Standard smoking cessation pamphlet
  Interventions: Behavioral: Standard smoking cessation intervention

INTERVENTIONS:
Behavioral: BTI — Brief Tobacco Intervention (BTI). The group intervention was designed to include the components of effective tobacco control programs for military personnel, and specifically tailored to the Technical Training environment. The intervention is approximately 40 minutes and delivered in a group format (e.g., groups of 50 Airmen). The format of the BTI is meant to be interactive, utilizing the Socratic teaching style and eliciting participation through the principles of motivational interviewing. A series of open-ended questions, reflections, and decisional balance, were used to increases motivation to remain tobacco free.
  Arms: BTI + Cigarette smoking military tailored pamphlet
Behavioral: Cigarette smoking military tailored pamphlet — The Airmen's Guide is 5×7 inches, 46 pages, with text and color illustration. The text covers the advantages of remaining tobacco-free after Basic Military Training, and the opportunity the ban provides to begin a lifetime without tobacco, focusing on cigarettes and smokeless tobacco. Information is included about challenges and coping suggestions for the times that Airmen are at particular risk of smoking. The text is supplemented by images created specifically for Airmen and designed to reinforce the messages that smoking: 1) is responsible for more fatalities than combat; 2) conveys a negative image to civilians; and 3) impedes military readiness and promotion through the ranks.
  Other Names: The Airman's Guide to Remaining Tobacco Free
  Arms: BTI + Cigarette smoking military tailored pamphlet; Cigarette smoking military tailored pamphlet
Behavioral: Standard smoking cessation intervention — This booklet is a 36-page, comprehensive guide for quitting smoking with 7 pages dedicated to relapse-prevention.
  Other Names: National Cancer Institute's Clearing the Air
  Arms: Standard smoking cessation pamphlet

SUMMARY:
While the military has taken steps to reduce tobacco use over the past two decades, over a quarter of new military recruits report regular tobacco use prior to enlistment. This rate is higher than the national prevalence of 21.3% of US adults. Brief health prevention programs may be particularly effective for Airmen in Technical Training, given that all Airmen have been tobacco free for 11 ½ weeks and nearly 2/3rds are confident that they won't return to tobacco. We have developed and validated a Brief Tobacco Intervention (BTI) that is currently being implemented as part of Technical Training. We found that a motivational interviewing based, 40 minute BTI was efficacious in increasing perceived harm and decreasing intentions to use tobacco in a sample of 1055 Air Force trainees. Although we obtained significant positive changes in latent cognitive constructs for tobacco behavior that are highly predictive of future tobacco use in youth and young adults, the Little et al study did not obtain measures of actual tobacco resumption following the ban on tobacco in Air Force training. Given that 69.8% of all tobacco resumption/initiation occurs in Technical Training, a study that evaluates the short-term impact of our BTI on actual tobacco use is necessary prior to conducting the full scale R01 that would evaluate the long term efficacy of the BTI intervention. Thus, we propose the following Specific Aims: (1) To recruit approximately 2,000 Air Force trainees at the beginning of Technical Training at Joint Base San Antonio-Lackland Air Force in San Antonio, Texas during the 11 ½ week involuntary cessation ban; (2) To randomize participants to either (a) receive our cigarette smoking military tailored pamphlet (HL095758), The Airmen's Guide to Remaining Tobacco Free (Airmen's Guide; which has been disseminated and is now the standard of care in the Air Force) or (b) the Airmen's Guide + Brief Tobacco Intervention (BTI); (3) To determine the short-term (3 month, end of Technical Training) efficacy of the intervention on tobacco abstinence. Our primary outcome is tobacco abstinence at the end of Technical Training to determine an estimated effect size as well as establish the requisite preliminary work for a subsequent R01. Given that over 220,000 new recruits enter the military annually in one of the service branches, the public health implications of an effective brief tobacco intervention targeting the most commonly used tobacco for military personnel in Technical Training is considerable. If the BTI is proven efficacious it can be easily disseminated to other service branches that have similar tobacco bans during Technical Training.

DETAILED DESCRIPTION:
This study builds on preliminary data from this population based on over 1,000 Airmen. We have developed and validated a Brief Tobacco Intervention (BTI) that is currently being implemented as part of Technical Training. We found that a motivational interviewing based, 40 minute BTI was efficacious in increasing perceived harm and decreasing intentions to use tobacco in a sample of 1055 Air Force trainees. Although we obtained significant positive changes that are predictive of future tobacco use in self-reported intent to use (decreased) and self-reported perceived harm (increased), we did not obtain measures of actual tobacco resumption following the tobacco use ban in Air Force training. This study will obtain and analyze data on these measures.

Airmen will be consented in the presence of an Ombudsman and randomly assigned to either (1) BTI + The Airman's Guide to Remaining Tobacco Free at the beginning of Technical Training, (2) The Airman's Guide to Remaining Tobacco Free (no BTI), or (3) the standard smoking cessation pamphlet (no BTI). All interventions in this study are command-directed interventions provided to all Technical Training students in the 37th Training Group. Airmen who are willing to participate in the study will be consented before the administration of the brief assessment of the BTI. Immediately following the intervention, consented Airmen will receive another assessment to evaluate any immediate changes in several important cognitive constructs (e.g., perceived harm, self-efficacy, perceived behavioral control, subjective norms, attitudes, intentions). At the end of Technical Training (3 months), consented Airmen will complete a final assessment to determine tobacco abstinence.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be Active duty Air Force Technical Training students from the 37th Training Group (JBSA Lackland), who are at least 18 years old.

Exclusion Criteria:

* Individuals unable to understand the consent procedures would be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2999 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
tobacco continuous abstinence | 3 months
  No tobacco use at 3 month follow-up since pre-assessment

CONTACTS AND LOCATIONS:
Locations (1):
- 37th Training Group, Lackland Air Force Base, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fahey MC, Talcott GW, McMurry TL, Klesges RC, Tubman D, Krukowski RA, Little MA. When, How, & Where Tobacco Initiation and Relapse Occur During U.S. Air Force Technical Training. Mil Med. 2020 Jun 8;185(5-6):e609-e615. doi: 10.1093/milmed/usaa016. PMID 32060547
- [Background] Little MA, Talcott GW, Bursac Z, Linde BD, Pagano LA, Messler EC, Ebbert JO, Klesges RC. Efficacy of a Brief Tobacco Intervention for Tobacco and Nicotine Containing Product Use in the US Air Force. Nicotine Tob Res. 2016 May;18(5):1142-9. doi: 10.1093/ntr/ntv242. Epub 2015 Oct 27. PMID 26508394
- [Result] Little MA, Fahey MC, Klesges RC, McMurry T, Talcott GW. Evaluating the Effects of a Brief Tobacco Intervention in the US Air Force. Nicotine Tob Res. 2020 Aug 24;22(9):1569-1577. doi: 10.1093/ntr/ntaa001. PMID 31903494